CLINICAL TRIAL: NCT03208556
Title: Pilot Study of Autologous Anti-CD19 4-1BB CAR T Cells With Cell-intrinsic PD1 Inhibition in Relapsed or Refractory B-cell Lymphoma
Brief Title: Safety and Efficacy of iPD1 CD19 eCAR T Cells in Relapsed or Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Marino Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhu, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017YJZ13
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-07

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPD1 CD19 eCAR T cells (Experimental): patients will receive a lymphodepletion chemotherapy prior to CAR T cell infusion
  Interventions: Biological: iPD1 CD19 eCAR T cells; Drug: Fludarabine and cyclophosphamide

INTERVENTIONS:
Biological: iPD1 CD19 eCAR T cells — iPD1 CD19 eCAR T cells are administrated in a 3-day split-dose regimen （d0, 30%; d1, 30%; d2, 40%）.
  CAR T cell dose escalation: 1×10^5 /kg，1×10^6 /kg，3×10^6 /kg，and 6×10^6 CAR T cells/kg
Drug: Fludarabine and cyclophosphamide — Fludarabine 25 mg/m2 d1-3; cyclophosphamide 250 mg/m2 d1-3. Lymphodepletion chemotherapy is completed 1 to 4 days before CAR T cell infusion

SUMMARY:
PD1 pathway is critical in determining the response to CAR T cell therapy. Emerging data suggested that Inhibition of PD1 could enhance the efficacy of CAR T cell therapy. iPD1 CD19 eCAR T cells is an enhanced version of the classical 2nd generation anti-CD19 4-1BB-costimulatory chimeric antigen receptor engineered T cells with cell-intrinsic PD1 inhibition by incorporation of a PD1 shRNA-expressing cassette in the CAR lentivector. This design will enhance the anti-tumor activities of CAR T cells by inhibiting PD1 induction after CAR T cell activation. This pilot, single arm, one center, dose-escalation, open label study is to determine the safety and efficacy of iPD1 CD19 eCAR T cells in relapsed or refractory CD19 positive lymphoma.

Subjects will be given a lymphodepletion chemotherapy comprised of Fludarabine and cyclophosphamide prior to CAR T cell infusion. The chemotherapy is completed 1 to 4 days before the first dost of iPD1 CD19 eCAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. CD19+ B cell lymphoma,verified by IHC or flow cytometry.
2. a prior history of at least one standard care of medication.
3. ineligible for allogeneic transplantation or relapsed after transplantation.
4. patients are 18 years older.
5. life expectancy > 3months.
6. ECOG ≤ 2.
7. satisfactory major organ functions: adequate heart function with LVEF≥50%; pulse oximetry of ≥ 90%; cockcroft-gault creatinine clearance≥40 ml/min; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3ULN; Bilirubin ≤2.0 mg/dl .
8. Blood: Hgb ≥ 80 g/L, ANC ≥ 1×10^9/L, PLT ≥ 50×10^9/L.
9. women of reproductive potential must have a negative pregnancy test. Male and female of reproductive potential must agree to use birth control during the study and one year post study.
10. measurable tumors.

Exclusion Criteria:

1. using immunosuppressive drugs or systemic steroids within one week of enrollment.
2. active infection.
3. HIV positive.
4. active hepatitis B virus infection or hepatitis C virus infection.
5. breastfeeding or pregnant women.
6. patients refuse to practice birth control during study and one year post study.
7. patients with a prior history of other malignances will be excluded from this study, but patients who have been cured from skin basal cell carcinoma or cervical cancer, or who have had their tumors removed by surgical resection but without further therapies and have more than 5 years of progression-free survival, can be included into the study.
8. currently enrolled in other study.
9. patients, in the opinion of investigators, may not be eligible or are not able to comply with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
safety of infusion of iPD1 CD19 eCAR T cells as assessed by the incidents of treatment related adverse events per NCI CTCAE V4.0 | 2 years
  incidents of treatment related adverse events per NCI CTCAE V4.0

SECONDARY OUTCOMES:
treatment response | 6 months
  The efficacy of infusion of iPD1 CD19 eCAR T cells is assessed according to the standardized response criteria for malignant lymphoma (Cheson BD, JCO, 2007), which is defined as complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD).
overall survival | 3 years
  Overall survival is defined as the time from receiving iPD1 CD19 eCAR T cells infusion to death for any cause.
progression-free survival | 2 years
  Progression-free survival (PFS) is defined as the time from receiving iPD1 CD19 eCAR T cell infusion to disease progression or death from any cause.

OTHER OUTCOMES:
Persistence of iPD1 CD19 eCAR T cells in patients | 2 years
  measured by quantitative PCR
proliferation of iPD1 CD19 eCAR T cells in patients | 6 months
  measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Zhitao Ying, MD, Study Director — Peking University Cancer Hospital & Institute; Xiaoyu Xiang, PhD, Study Director — Marino Biotechnology Co., Ltd.
Locations (1):
- Beijing Cancer Hosptical, Beijing, China